CLINICAL TRIAL: NCT00893256
Title: Prospective Double-Blind Randomized Comparison Study of Improvement in Negative Symptoms With Risperidone vs Risperidone +Citalopram Combination Therapy in Schizophrenia--a Clinical Study
Brief Title: Effect of Add-on Citalopram to Risperidone on Negative Symptoms in Schizophrenia
Acronym: RIS-CIT-SCH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Mental Health and Neuro Sciences, India (Other)
Responsible Party: Dean, NIMHANS
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NFRPA/006/2004
Record Dates: First submitted 2009-05-04; First posted 2009-05-05 (Estimated); Last update posted 2009-05-05 (Estimated); Status verified 2009-05

CONDITIONS: Schizophrenia; Negative Symptoms
Keywords: schizophrenia; risperidone; citalopram; secondary negative symptoms
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; Citalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Risperidone and citalopram (Experimental): 24 patients were randomized to receive add-on citalopram (20 mg/day) in a double-blind fashion to open-label risperidone (4-8 mg/day)
  Interventions: Drug: Risperidone; Drug: Citalopram
- Risperidone and placebo (Placebo Comparator): 24 patients were randomized to receive add-on placebo in a double-blind fashion to open-label treatment with risperidone (4-8 mg/day)
  Interventions: Drug: risperidone; Drug: Placebo

INTERVENTIONS:
Drug: Risperidone — Risperidone: tablet; oral; 4-6 mg/day; once daily; 12 weeks
  Other Names: Respidon
  Arms: Risperidone and citalopram
Drug: risperidone — Risperidone: tablet; 4-8 mg/day; once daily; 12 weeks
  Other Names: Respidon
  Arms: Risperidone and placebo
Drug: Citalopram — Citalopram: tablet; oral; 20 mg/day; once daily; 12 weeks
  Other Names: Citopam
  Arms: Risperidone and citalopram
Drug: Placebo — Placebo: once daily
  Arms: Risperidone and placebo

SUMMARY:
Negative symptoms in schizophrenia present a challenge to the clinician owing to their poorer response to conventional treatment with antipsychotics. Negative symptoms in schizophrenia may be secondary to psychotic symptoms, depressive symptoms, drug-related side effects or lack of environmental stimulation. Alternately, they may represent core features of the illness, characterized as primary deficit symptoms. Previous studies have suggested that atypical antipsychotics may be beneficial in improving deficit symptoms of schizophrenia. This study aimed at characterizing the nature of improvement of negative symptoms in the early phase (12 weeks) of treatment with the atypical antipsychotic, risperidone. In order to account for factors contributing to improvement in secondary negative symptoms, ratings were carried out of change in positive symptoms, depressive symptoms and drug-related side effects. Further, add-on citalopram or placebo were administered in a double-blind design to study the effect of selective serotonin reuptake inhibitor (SSRI) augmentation of risperidone on negative symptoms. The investigators hypothesized that the improvement in negative symptoms during the initial phase (12 weeks) of treatment with risperidone will be largely accounted for by improvement in secondary negative symptoms, rather than of the primary deficit symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling DSMIV Criteria for Schizophrenia
* The patient should be drug naïve or drug free for one month (oral antipsychotic) or three months of parental antipsychotic
* Duration from onset < 5 years
* Informed consent

Exclusion Criteria:

* Patient with any other current Axis I or Axis II comorbid disorders
* Comorbid substance abuse or dependence except nicotine or caffeine
* Presence of significant medical disorder such as epilepsy, uncontrolled hypertension and diabetes mellitus, thyroid disorder
* Patient who has not responded to adequate course of risperidone (with reference to dose and duration)
* Treatment-resistant schizophrenia defined as non-response to three different antipsychotics belonging to at least two different classes, one of which is an atypical agent and one of which is a depot neuroleptic
* Patient who has received ECT in past 3 months

Ages: 17 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2004-12; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Change in PANSS negative symptom score | 12 weeks

SECONDARY OUTCOMES:
Change in PANSS total score | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John P John, M.D., Principal Investigator — National Institute of Mental Health and Neurosciences, Bangalore, INDIA
Locations (1):
- National Institute of Mental Health and Neurosciences (NIMHANS), Bangalore, Karnataka, India